CLINICAL TRIAL: NCT00287651
Title: Effects of Pulsatile IV Insulin Delivery on Diabetic Retinopathy
Brief Title: Effects of Pulsatile IV Insulin Delivery on Diabetic Retinopathy in Patients With Types 1 and 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other); Global Infusions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H09-06; MH42900 and MH01386
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, With Complications
Keywords: Pulsatile intravenous insulin; Oral carbohydrate loading; Respiratory Quotients; Hypoglycemia
MeSH Terms: conditions — Diabetes Complications; Hypoglycemia | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Patients with diagnosed Diabetic Retinopathy are enrolled as treated with pulsatile intravenous insulin or as a control patient with weekly treatment sessions. Baseline and quarterly fundus photography is performed to measure and monitor progress.
  Interventions: Procedure: Pulsatile IV Insulin; Procedure: Effects of Pulsatile IV Insulin on Diabetic Retinopathy
- 1 (No Intervention): Patients diagnosed with Diabetic Retinopathy are enrolled as control patients that do not receive the pulsatile intravenous insulin therapy. Control patients come into the center receive baseline fundus photography and quarterly fundus photography to measure progress and outcomes of diabetic retinopathy and are compared to the patients who receive pulsatile intravenous insulin therapy.

INTERVENTIONS:
Procedure: Pulsatile IV Insulin — Intravenous Insulin is provided in a pulsed manner based upon weekly physician orders the amount of insulin provided is dependent on patients level of insulin resistance.
  Arms: 2
Procedure: Effects of Pulsatile IV Insulin on Diabetic Retinopathy — Control Patients are not given pulsatile intravenous insulin therapy during the study.
  Arms: 2
Procedure: Effects of Pulsatile IV Insulin on Diabetic Retinopathy — Intravenous Insulin is provided in a pulsed manner based upon weekly physician orders the amount of insulin provided is dependent on patients level of insulin resistance.
  Other Names: Humilin, Humolog, Novolog, Epidra
  Arms: 2

SUMMARY:
Diabetic Retinopathy is the leading cause of blindness in the world. Previous studies have documented beneficial effects of physiologic administration of pulsatile insulin on a variety of diabetic complications such as nephropathy, hypertension, glycemic control, etc. Similar pathogenetic mechanisms have been postulated for diabetic retinal disease. This study examines the effect of pulsatile insulin on patients with varying stages of diabetic retinal disease.

DETAILED DESCRIPTION:
Diabetic retinopathy is one of the leading causes of blindness in the world. Signs of retinopathy are detected in almost 100% of type 1 diabetic patients who have had their disease for at least 20 years and almost 100% of type 2 diabetic patients with the similar duration of disease (1). Histopathologic findings range from microaneurysms and cotton wool spots to more ominous neovascularization. The latter process, known as proliferative diabetic retinopathy, can progress to total blindness if untreated. The biochemical mechanisms responsible for PDR have been extensively studied, and appear to be multifactorial. Associated findings include abnormalities of vasoactive peptides such as vascular endothelial growth factor (VEGF), pigment epithelium derived factor (PEDF), and insulin-like growth factor (ILF-1), lipids, oxidative pathways, enzymatic pathways, such as protein kinase, and carbohydrate metabolism (1-4). Whether these (and other) factors are interrelated or have a common underlying defect is unknown. The common endpoint, however, is vascular leakage with neovascularization. Current therapeutic regimens based on these biochemical abnormalities have to date been unsuccessful in stemming the progression of proliferative diabetic retinopathy. Current treatment strategies emphasize glycemic and blood pressure control, with laser photocoagulation and vitrectomy for advanced cases (5).

Early retinal disease in diabetic patients may take the form of diabetic macular edema (DME). This is observed in 20% to 25% of both type 1 and type 2 diabetic patients. The pathophysiology of DME involves the leakage of plasma from small vessels in the macula. Resorption of this fluid followed by hard exudate formation can lead to severe impairment of central vision (6).

Anecdotal evidence from ophthalmologic institutions (Houston Eye Institute, Shands at University of Florida, Bascom Palmer Eye Institute) suggests that this treatment arrests the progression of retinal disease in patients with proliferative diabetic retinopathy. The mechanism of this effect is unknown, but may be related to reversal of retinal ischemia or downregulation of vasoactive peptides by restoration of hepatic metabolism.

Protocol

This study is designed as a prospective, controlled, single blinded evaluation of pulsatile insulin in the role of diabetic retinopathy. The patients entered into the study will be from two distinct sources. First, in conjunction with a national eye imaging company, patients with known type 1 or type 2 diabetes will be evaluated for retinal disease. This evaluation will consist of mydriatic fundus photography in diabetic patients not having had recent ophthalmologic evaluation (period greater than 12 months). The fundus photographs will be read by an observer under the auspices of the Wilmer Ophthalmologic Institute at Johns Hopkins Hospital. Classifications of patients will be evaluated in this study include:

I Patients with non high risk proliferative diabetic retinopathy II Patients with severe non proliferative diabetic retinopathy

Patients who are diagnosed as one of these classifications will be offered entrance into the study. Study patients will be matched for age, sex, and disease severity into a treatment and control group. All study patients will be evaluated in conjunction with an ophthalmologist. This evaluation will include clinical examination and fundus photography. Treatment group patients will undergo weekly pulsatile insulin delivery sessions as per protocol above. Control group patients will have weekly clinic visits to maximize glycemic and hypertensive control. All patients will repeat their fundus photography at three month intervals, with ophthalmologic evaluation as above every six months, or more often if requested by the ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* We will include up to 500 patients both male and female over the age of 18 diagnosed with type 1 or type 2 diabetes mellitus.
* All patients must be diagnosed with type 1 or type 2 diabetes.
* Fundus photographs will be examined by an independent retinal specialist and the patients will be stratified into the three groups as outlined above.
* Endocrinologist must assess and approve patient for participation in this study
* Patient must have the ability to swallow without difficulty and ability to commit to the weekly time requirements associated with the study.

Exclusion Criteria:

* Other causes of complications not related to diabetes
* Lack of intravenous access
* Pregnancy
* Alcohol abuse, drug addiction or the use of illegal drugs
* Positive HIV
* Inability to breathe into metabolic measurement cart for respiratory quotients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Serial fundus photography | Stabilization of retinal blood vessel degeneration

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, Ph.D, Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University Center for Complex Systems and Brain Sciences, Boca Raton, Florida, United States

REFERENCES:
- [Background] Frank RN. Diabetic retinopathy. N Engl J Med. 2004 Jan 1;350(1):48-58. doi: 10.1056/NEJMra021678. No abstract available. PMID 14702427
- [Background] Caldwell RB, Bartoli M, Behzadian MA, El-Remessy AE, Al-Shabrawey M, Platt DH, Caldwell RW. Vascular endothelial growth factor and diabetic retinopathy: pathophysiological mechanisms and treatment perspectives. Diabetes Metab Res Rev. 2003 Nov-Dec;19(6):442-55. doi: 10.1002/dmrr.415. PMID 14648803
- [Background] Singleton JR, Smith AG, Russell JW, Feldman EL. Microvascular complications of impaired glucose tolerance. Diabetes. 2003 Dec;52(12):2867-73. doi: 10.2337/diabetes.52.12.2867. PMID 14633845
- [Background] Misra A, Kumar S, Kishore Vikram N, Kumar A. The role of lipids in the development of diabetic microvascular complications: implications for therapy. Am J Cardiovasc Drugs. 2003;3(5):325-38. doi: 10.2165/00129784-200303050-00004. PMID 14728067
- [Background] Jain A, Sarraf D, Fong D. Preventing diabetic retinopathy through control of systemic factors. Curr Opin Ophthalmol. 2003 Dec;14(6):389-94. doi: 10.1097/00055735-200312000-00012. PMID 14615645
- [Background] Fong DS, Aiello L, Gardner TW, King GL, Blankenship G, Cavallerano JD, Ferris FL 3rd, Klein R; American Diabetes Association. Diabetic retinopathy. Diabetes Care. 2003 Jan;26 Suppl 1:S99-S102. doi: 10.2337/diacare.26.2007.s99. No abstract available. PMID 12502630